CLINICAL TRIAL: NCT02083978
Title: Neuromorphometry of Psychosis in Bipolar Disorder
Brief Title: Bipolar Research Study Using MR Imaging
Status: Completed | Type: Observational
Sponsor: Washington University Early Recognition Center (Other)
Responsible Party: Sponsor
Other Study IDs: 201105453
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Bipolar Affective Disorder
Keywords: Bipolar Disorder; Magnetic Resonance Imaging (MRI) scanning
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bipolar Diagnosis: Individuals identified as having a Bipolar Diagnosis with a manic episode
  Interventions: Other: MRI scanning
- Control: Individuals identified as not having a major psychiatric diagnosis
  Interventions: Other: MRI scanning

INTERVENTIONS:
Other: MRI scanning

SUMMARY:
In this proposal, the investigators will focus on subcortical gray and white matter structures commonly found to be abnormal in schizophrenia. Thus, the investigators will evaluate the volume and shape of the hippocampus, thalamus and basal ganglia, as well as measures of structural integrity of the corpus callosum and its various subregions.

DETAILED DESCRIPTION:
There are relatively few studies evaluating brain structure in bipolar disorder (BD), the results of which have been largely inconsistent, both in terms of what abnormalities are present in BD and whether they show any similar abnormalities to those found in schizophrenia. One possibility that might explain the varying degree of reported similarity in structural findings in schizophrenia and BD is that there might be effects of BPD diagnostic subtype associated with brain structure. One viewpoint that contrasts schizophrenia and BD considers psychotic (PBD) to differ from non-psychotic (NPBD) subtypes in terms of shared pathophysiology with schizophrenia. PBD has been reported as being of special interest, as it shares symptomatic overlap with schizophrenia, "runs in families", shares a chromosomal linkage to the 13q13-32 and 22q12 with schizophrenia, shows similar increases in dopamine receptor Bmax induced by [c-11] N-methylspiperone positron emission tomography and similar working memory impairments as in schizophrenia. If PBP and NPBP are associated with different forms of brain pathology, then merging the two entities into a single "bipolar group" might obscure relevant anatomic differences if these occur primarily in only one group. In this proposal, the investigators will focus on subcortical gray and white matter structures commonly found to be abnormal in schizophrenia. Thus, the investigators will evaluate the volume and shape of the hippocampus, thalamus and basal ganglia, as well as measures of structural integrity of the corpus callosum and its various subregions.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-30
* diagnosed with Bipolar Disorder

Exclusion Criteria:

* history of head injury
* unstable medical condition

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2010-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
subcortical grey and white matter structures | within one month of study enrollment
  Evaluation of the volume and shape of the hippocampus, thalamus and basal ganglia, as well as measures of structural integrity of the corpus callosum and its various subregions.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Mamah, M.D, MPE, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States